CLINICAL TRIAL: NCT07264075
Title: A Randomized, Open-label, Multicenter, Phase 3 Trial of Ivonescimab Alone or With Ligufalimab Versus Pembrolizumab in First-line Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Study Comparing Ivonescimab Alone or Ivonescimab in Combination With Ligufalimab Versus Pembrolizumab for the Treatment of SCCHN
Acronym: ILLUMINE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Akeso Biopharma Co., Ltd. (Unknown); Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2024-04; 2025-522996-27-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-29; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma Head and Neck Cancer (HNSCC)
Keywords: first-line recurrent and/or metastatic
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bras A: Ivonescimab (Experimental): Ivonescimab (10 mg/kg iv, 60 min ± 10 min infusion, Q3W)
  Interventions: Drug: Ivonescimab 10 mg/kg
- Bras B: Ivonescimab - Ligufalimab (Experimental): Ivonescimab (10 mg/kg iv, 60 min ± 10 min infusion, Q3W), and ligufalimab (45 mg/kg iv, 120 min ± 15 min infusion, Q3W).
  Interventions: Drug: Ivonescimab 10 mg/kg; Drug: Ligufalimab
- Bras C: Pembrolizumab (Active Comparator): Pembrolizumab (200 mg iv, 60 min ± 10 min infusion, Q3W).
  Interventions: Drug: Pembrolizumab (KEYTRUDA ®)

INTERVENTIONS:
Drug: Ivonescimab 10 mg/kg — Ivonescimab is a humanized immunoglobulin (Ig) G1 monoclonal antibody (mAb) being investigated as a cancer immunotherapy agent. Ivonescimab binds to human VEGF-A which is involved in tumor angiogenesis, and to human PD-1 that is a cell surface receptor expressed primarily on activated T cells and acts to inhibit T cell activation.
  Other Names: AK112
  Arms: Bras A: Ivonescimab; Bras B: Ivonescimab - Ligufalimab
Drug: Ligufalimab — AK117 is a humanized IgG4 mAb being investigated as a cancer immunotherapy agent
  Other Names: AK117
  Arms: Bras B: Ivonescimab - Ligufalimab
Drug: Pembrolizumab (KEYTRUDA ®) — Pembrolizumab is a humanized monoclonal antibody (IgG4 kappa isotype with stabilizing sequence alteration in the Fc region) against PD-1 (programmed cell death-1), produced in Chinese hamster ovary cells by recombinant DNA technology.
  Other Names: Keytruda
  Arms: Bras C: Pembrolizumab

SUMMARY:
This is a randomized, open-label, active-comparator-controlled, multi-regional, three-arm, phase 3 study comparing the efficacy and safety of ivonescimab in combination with ligufalimab to pembrolizumab and of ivonescimab alone to pembrolizumab as first-line treatment in patients with recurrent or metastatic (R/M) PD-L1-positive squamous cell carcinoma of the head and neck (HNSCC).

The objective of this study is to improve first-line survival in patients with recurrent or metastatic PD-L1-positive HNSCC (CPS ≥ 1). Overall survival (OS) was chosen as the primary endpoint.

Patients will receive the following treatment regimens in accordance with the study treatment plan until disease progression, death, intolerable toxicity, or the occurrence of another protocol-specified treatment discontinuation criterion, whichever occurs first.

* ARM A: Ivonescimab (10 mg/kg iv, 60 min ± 10 min infusion, Q3W)
* ARM B: Ivonescimab (10 mg/kg iv, 60 min ± 10 min infusion, Q3W), and ligufalimab (45 mg/kg iv, 120 min ± 15 min infusion, Q3W).
* ARM C (control arm): Pembrolizumab (200 mg iv, 60 min ± 10 min infusion, Q3W). The total duration of treatment is up to 24 months

ELIGIBILITY:
Inclusion Criteria:

1. Patient capable of voluntary giving her/his written informed consent.
2. Age ≥ 18 and < 80 years old at the time of enrolment.
3. Eastern Cooperative Oncology Organization (ECOG) performance status score of 0 or 1.
4. Expected survival ≥ 6 months at randomization.
5. Patient is histologically and/or cytologically confirmed to have r/m HNSCC (according to the International Union Against Cancer and the American Joint Committee on Cancer 8th edition staging system) with a primary tumour initially or currently located in the oral cavity, oropharynx, hypopharynx, or larynx.
6. HPV status test results based on tumour tissue samples must be obtained prior to randomization for patients with oropharyngeal cancer.
7. No prior systemic anti-tumour therapy for R/M HNSCC. Note: Patients who have previously received adjuvant/neoadjuvant chemotherapy with curative intent for non-metastatic disease, radiotherapy, or radical radiotherapy in combination with chemotherapy or cetuximab/EGFR based therapy for locally advanced disease are eligible for this study if disease progression occurs > 6 months after the end of the last treatment.
8. At least one measurable lesion according to RECIST v1.1, or measurable lesion with clear radiographic progression after local therapy, and the lesion must be suitable for repeated accurate measurements (see Appendix 3).
9. Tumours must be PD-L1 positive (CPS ≥ 1) as confirmed by CE-IVD immunohistochemistry assay based on local assessment with any assay validated for HNSCC in a laboratory compliant with National provisions. The measurement of PD-L1 protein expression can be performed based on archival tissue sample before the diagnosis of R/M tumour or based on tissue sample obtained after the diagnosis of a R/M tumour.
10. Good organ function is determined by the following requirements:

    a.Haematology (satisfactory laboratory test results obtained during the screening period, and no blood components used within 14 days of cell growth factor supportive therapy): i.Absolute neutrophil value (ANC) ≥ 1.5×109/L (1,500/mm3) ii.Platelet count ≥ 100×109/L (100,000/mm3) iii.Haemoglobin ≥ 10 g/dL b.Kidneys: i.Calculated creatinine clearance (Appendix 4) ≥ 50 mL/min ii.Urine protein ≤ 2+ or 24 hours (h) urine protein quantification < 1.0 g c.Liver: i.Serum total bilirubin ≤ 1.5× upper limit of normal (ULN); for patients with liver metastases or confirmed/suspected Gilbert syndrome, ≤ 3 × ULN ii.AST and ALT ≤ 2.5×ULN; For patients with liver metastases, AST and ALT ≤ 5×ULN iii.Serum albumin ≥ 28 g/L d.Coagulation function: International normalized ratio (INR) and/or activated partial thromboplastin time (APTT) ≤ 1.5× ULN. This applies only to patients who are not on therapeutic anti- coagulation. Patients receiving therapeutic anti-coagulation should be on a stable dose.

Exclusion Criteria:

1. Primary tumour site (any histology) of nasopharynx, nasal cavity, sinuses, salivary glands, thyroid or parathyroid glands, skin, or unknown primary site of tissue origin.
2. Patient with malignancies other than HNSCC within 3 years prior to enrolment. Patients with other tumours that have been cured through local treatment, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ, are not excluded.
3. Concurrent enrolment in another clinical study, unless it is an observational, non-interventional clinical study or a follow-up period of an interventional study; Received study treatment within 4 weeks prior to randomization.
4. Prior treatment with systemic anti-angiogenic drugs.
5. Previous head and neck re-irradiation for recurrent/metastatic disease
6. Prior immunotherapy, including immune checkpoint inhibitors (e.g., anti-PD-1/L1 antibody, anti- CTLA-4 antibody, anti-TIGIT antibody, anti-LAG3 antibody, anti-CD47, anti-SIRPα, etc.), immune checkpoint agonists (e.g., ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), immune cell therapy, and any other treatment that targets tumour immunity including therapeutic tumour vaccine, and other adjuvant/neoadjuvant anti-PD-1 based therapy.
7. Patients with ulcers on the skin surface related to the current cancer during the screening period, superficial or protruding skin lesions with excessive surface tension and a greater risk of ulceration, or other patients with a greater risk of ulceration as assessed by the investigator. Patients with recent tracheostomy involving the tumour which are at risk of bleeding.
8. Imaging during the screening period shows that the tumour invades/infiltrates the surrounding important organs (such as trachea, oesophagus, and based on investigator assessment ofbleeding risk) and/or large blood vessels in the neck (such as subclavian artery, common internal and/or external carotid artery, etc.) or if the investigator judges that entering the study might cause a potential risk of bleeding.
9. Presence of brainstem, meningeal metastases, spinal cord metastases or compression, or leptomeningeal disease.
10. Received curative head and neck radiotherapy within 6 months prior to randomization. Palliative local treatment for non-head and neck areas carried out within 3 weeks before randomization; Received non-specific immunomodulatory therapy (such as interleukin, interferon, thymus peptide, tumour necrosis factor, etc.) within 2 weeks prior to randomization, excluding IL-11 for the treatment of thrombocytopenia.
11. Presence of active autoimmune disease requiring systemic therapy (e.g., treatment with disease-modifying drugs, corticosteroids, immunosuppressants) within 2 years prior to randomization. Alternative therapies (e.g., thyroxine, insulin, or those targeting the adrenal glands or pituitary) and physiologic corticosteroid replacement therapy for pituitary insufficiency are not considered systemic treatment.
12. History of immunodeficiency; Those who have history of positive test for HIV antibodies; Current long-term use of systemic corticosteroids or other immunosuppressants is excluded.
13. Previous or current non-infectious pneumonitis/interstitial lung disease requiring systemic glucocorticoid therapy, or current presence of lung diseases including but not limited to the following: pneumoconiosis, silicosis, drug-related pneumonia, pulmonary diseases with severe impairment of lung function, etc.
14. Severe infection within 4 weeks prior to randomization, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; Active non-severe infection that has received systemic anti-infective therapy within 2 weeks prior to randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization to the date of death from any cause up to 54 months
  the time from the date of randomization to the date of death from any cause. Patients still alive at the time of analysis will be censored at the date of their last known alive date

IPD SHARING:
Plan to Share IPD: Yes
The study will be conducted in Europe and China, with GORTEC as the sponsor. A single, secure database will be used, and pseudonymized participant data will be shared among the partners.